CLINICAL TRIAL: NCT06255015
Title: Breastfeeding Planning Card Feasibility Study
Brief Title: Breastfeeding Planning Card Trial in Scotland
Acronym: CARRDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stirling (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Principal Investigator, David Comerford, Professor of Behavioural Science, University of Stirling
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IRAS: 316125
Record Dates: First submitted 2023-03-28; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A regression discontinuity design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding toolkit card (Active Comparator): 50% of participants will be allocated to the intervention group, and receive a breastfeeding toolkit card at the 24 week appointment.
  The Breastfeeding toolkit provides advice on circumventing common breastfeeding problems and contact details for breastfeeding support services.
  Interventions: Device: Breastfeeding toolkit card
- No planning card (No Intervention): 50% of women will receive routine antenatal care only.

INTERVENTIONS:
Device: Breastfeeding toolkit card — The card is delivered at 24 weeks and is also referred to in the 32 and 36 week antenatal meetings. It will also be referred to in the first 24 hours post-partum and in home visits.
  Arms: Breastfeeding toolkit card

SUMMARY:
This study evaluates the efficacy of a "breastfeeding toolkit" card delivered as part of antenatal care in promoting breastfeeding maintenance.

DETAILED DESCRIPTION:
The project is an evaluation of an intervention that will start on January 1 2024.

From January 1 2024 through to March 31st 2024 midwives will present to patients attending their 24 week antenatal appointment a breastfeeding toolkit card.

The trial compares breastfeeding rates across patients who receive the card and those whose 24-week antenatal appointment occurred in the three months October 1 2023 - December 31 2023.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in NHS Grampian

Exclusion Criteria:

None

Min Age: 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women in NHS Grampian
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
breastfeeding rates at 6-8 weeks post-partum | 6-8 weeks
  Proportion of women recorded as breastfeeding by their home visitor at 6-8 weeks post-partum

SECONDARY OUTCOMES:
breastfeeding rates at 10-14 days post-partum | 10-14 days
  Proportion of women recorded as breastfeeding by their home visitor at 10-14 days post-partum

CONTACTS AND LOCATIONS:
Overall Officials: David Comerford, Principal Investigator — Stirling University
Locations (1):
- University of Stirling, Stirling, Stirlingshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No